CLINICAL TRIAL: NCT02424708
Title: Phase IIb Study of Intranasal Glutathione in Parkinson's Disease
Acronym: (in)GSH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bastyr University (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 14-1443
Record Dates: First submitted 2015-04-15; First posted 2015-04-23 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Parkinson's Disease
Keywords: Reduced Glutathione; Intranasal; (in)GSH; Parkinson's Disease; Glutathione; Uptake; central nervous system
MeSH Terms: conditions — Parkinson Disease | interventions — Glutathione; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): The study medication is packaged in sterile 1 ml pre-filled syringes, containing saline, which will be delivered intranasally.
  Interventions: Drug: Placebo
- Reduced Glutathione 100mg (Active Comparator): The study medication is packaged in sterile 1 ml pre-filled syringes, containing 100 mg/ml of reduced glutathione (GSH), which will be delivered intranasally.
  Interventions: Drug: Reduced Glutathione 100mg
- Reduced Glutathione 200mg (Active Comparator): The study medication is packaged in sterile 1 ml pre-filled syringes, containing 200 mg/ml of reduced glutathione (GSH), which will be delivered intranasally.
  Interventions: Drug: Reduced Glutathione 200mg

INTERVENTIONS:
Drug: Reduced Glutathione 100mg — 100mg GSH delivered intranasally, three times a day for 12 weeks, in 1 cc sterile saline using a syringe with a Mucosal Atomization Device (MAD) tip.
  Other Names: (in)GSH
  Arms: Reduced Glutathione 100mg
Drug: Reduced Glutathione 200mg — 200mg GSH delivered intranasally, three times a day for 12 weeks, in 1 cc sterile saline using a syringe with a Mucosal Atomization Device (MAD) tip.
  Other Names: (in)GSH
  Arms: Reduced Glutathione 200mg
Drug: Placebo — Saline delivered intranasally, three times a day for 12 weeks, in 1 cc sterile saline using a syringe with a Mucosal Atomization Device (MAD) tip.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Glutathione is an important nutrient for brain function and loss of glutathione has been implicated in Parkinson's disease. Glutathione is an antioxidant made in the body out of three amino acids, the nutrients that make up protein. This study will determine whether administration of either dose of glutathione, as a nasal spray, improves PD symptoms over time in a population of individuals with Parkinson's disease (PD).

DETAILED DESCRIPTION:
The study begins with a pre-screening telephone interview. During this conversation participants will be asked a series of questions that will help us identify whether they are eligible for participation in this study. The pre-screening interview process will take approximately 10 minutes and will include all screening criteria that does not require clinical or laboratory examination

All routine research visits will take place at Bastyr University Campus (Kenmore, WA). Participants will be asked to schedule visits at approximately the same time of day each visit .If they are on medications, we would like them to take their medications as they normally would on the day of the visit. Participants will be randomly assigned to one of three different study groups- a low dose group, a high dose group, or a placebo group.

Study participants will invited to volunteer for two magnetic resonance imagine (MRI) scans as part of this study, an optional part of study participation. For those who volunteer and qualify, MRIs will be performed at the University of Washington Radiology Department early in the morning. One scan will be taken at baseline before taking glutathione and the second upon completion of the study medication. There will be a separate consent form for those who participate in the imaging portion of this study. Among the participants who volunteer, the first 15 to qualify for an MRI scan will be scheduled according to MRI availability.

If participants are enrolled in the study, they will be asked to keep a daily log of actual frequency of administration of study medication, if any, as well as any changes in their PD symptoms, any adverse events they might experience, and their general well-being. We are giving participants enough medication to last four weeks, until the date of their next appointment. The medication should be taken three times a day (morning, afternoon, and evening).

Visit 1- Baseline: (Approximately 1 hour)

* Urine sample
* Venipuncture (blood draw, (40 mL / ~3 Tbsp) to assess blood antioxidant status..
* Clinical assessment of PD severity: Unified Parkinson's Disease Rating Scale (UPDRS), which involves assessing degree of tremor, ability to walk across the room, questions about ability to function independently (i.e. button your own shirt, feed yourself), and questions about mental health, including depression and intellectual impairment.
* Participant will be taught how and when to administer the study medication and be given a 1-month supply.

Visit 2- Week 4 follow-up: (Approximately 1 hour)

* Urine sample
* Venipuncture (blood draw, (40 mL / ~3 Tbsp) to assess blood antioxidant status..
* Clinical assessment of PD severity: Unified Parkinson's Disease Rating Scale (UPDRS) and Webster-Step Second test involve assessing degree of tremor, ability to walk across the room, questions about ability to function independently (i.e. button your own shirt, feed yourself), and questions about mental health, including depression and intellectual impairment.
* Participant will be asked to return any unused study medication and applicator tips from the first month of the study and be given the next 1-month supply.
* We will inquire about medication changes and collect medication use logs.

Visit 3- Week 8 follow-up: (Approximately 1/2 hour)

* Participant will be asked to return any unused study medication from the second month of the study and be given the next 1-month supply.
* We will inquire about medication changes and collect medication use logs.

Visit 4- Week 12 follow-up: (Approximately 1 hour)

* Urine sample
* Venipuncture (blood draw, (40 mL / ~3 Tbsp) to assess blood antioxidant status..
* Clinical assessment of PD severity: Unified Parkinson's Disease Rating Scale (UPDRS) to assess degree of tremor, ability to walk across the room, questions about ability to function independently (i.e. button your own shirt, feed yourself), and questions about mental health, including depression and intellectual impairment.
* Participants will be asked to return any unused study medication from the third month of the study.
* We will inquire about medication changes and collect medication use logs.

Visit 5- Week 16 follow-up: (Approximately 1 hour)

This visit is included to determine whether there are any lasting effects of the study medication one month following discontinuation of use. The visit will include:

* Urine sample
* Venipuncture (blood draw, (40 mL / ~3 Tbsp) to assess blood antioxidant status..
* Clinical assessment of PD severity: Unified Parkinson's Disease Rating Scale (UPDRS) which involves assessing degree of tremor, ability to walk across the room, questions about ability to function independently (i.e. button your own shirt, feed yourself), and questions about mental health, including depression and intellectual impairment.

Overall, approximately 5 hours will be required for study participation. Blood draws will occur at most, but not all visits, and will not exceed 4 Tbsp per month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD made by a clinical neurologist within the previous 10 years
* A modified Hoehn & Yahr Stage <3
* Age >21
* Subjects must be able to attend study visits at baseline, weeks 4, 8, 12, and 16.
* Subjects must be able to demonstrate, or have a caregiver administer, medication.
* Dose and frequency of pharmaceutical medications must be stable for 1 month prior to enrollment.
* Dose and frequency of naturopathic medications must be stable for 1 month prior to enrollment.
* Diet, exercise, and medications must be kept constant throughout participation in the study. (Medication changes considered essential by a participant's physician will be permitted and recorded).
* Ability to read and speak English.
* MRI cohort: Additional inclusion criteria specific to MRI.

Exclusion Criteria:

* Dementia as evidenced by a Montreal Cognitive Assessment score of less than 24.
* Diseases with features common to PD (e.g., essential tremor, multiple system atrophy, progressive supranuclear palsy)
* Epilepsy
* A history of stroke
* The presence of other serious illnesses
* Respiratory disease (e.g. asthma, COPD)
* A history of brain surgery
* A history of structural brain disease
* A history of intranasal telangiectasia
* Supplementation with glutathione, and agents shown to increase glutathione, will not be permitted and their use will necessitate a 90-day washout period; this will be required for all forms of glutathione and the glutathione precursor, N-acetylcysteine.
* Pregnant or at risk of becoming pregnant (i.e., unwilling to use birth control if a sexually active, pre-menopausal female). Urine pregnancy tests will be administered to pre-menopausal women.
* MRI cohort: Additional exclusion criteria specific to MRI.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Unified Parkinson's Disease Rating Scale (UPDRS) Score | 12 weeks

SECONDARY OUTCOMES:
Red blood cell (RBC) GSH levels will be measured at baseline, week 4, week 12, and 16. | up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laurie K Mischley, NDMPHPhD(c), Principal Investigator — Bastyr University
Locations (2):
- United States (2):
  - Bastyr University, Kenmore, Washington
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Allen J. Inhaled glutathione for the prevention of air pollution-related health effects: a brief review. Altern Ther Health Med. 2008 May-Jun;14(3):42-4. PMID 18517105
- [Background] Baker MA, Cerniglia GJ, Zaman A. Microtiter plate assay for the measurement of glutathione and glutathione disulfide in large numbers of biological samples. Anal Biochem. 1990 Nov 1;190(2):360-5. doi: 10.1016/0003-2697(90)90208-q. PMID 2291479
- [Background] Chinta SJ, Andersen JK. Reversible inhibition of mitochondrial complex I activity following chronic dopaminergic glutathione depletion in vitro: implications for Parkinson's disease. Free Radic Biol Med. 2006 Nov 1;41(9):1442-8. doi: 10.1016/j.freeradbiomed.2006.08.002. Epub 2006 Aug 7. PMID 17023271
- [Background] Dexter DT, Sian J, Rose S, Hindmarsh JG, Mann VM, Cooper JM, Wells FR, Daniel SE, Lees AJ, Schapira AH, et al. Indices of oxidative stress and mitochondrial function in individuals with incidental Lewy body disease. Ann Neurol. 1994 Jan;35(1):38-44. doi: 10.1002/ana.410350107. PMID 8285590
- [Background] Eyer P, Podhradsky D. Evaluation of the micromethod for determination of glutathione using enzymatic cycling and Ellman's reagent. Anal Biochem. 1986 Feb 15;153(1):57-66. doi: 10.1016/0003-2697(86)90061-8. PMID 3963383
- [Background] Schapira AH. Progress in neuroprotection in Parkinson's disease. Eur J Neurol. 2008 Apr;15 Suppl 1:5-13. doi: 10.1111/j.1468-1331.2008.02055.x. PMID 18353131
- [Background] Schulz JB, Lindenau J, Seyfried J, Dichgans J. Glutathione, oxidative stress and neurodegeneration. Eur J Biochem. 2000 Aug;267(16):4904-11. doi: 10.1046/j.1432-1327.2000.01595.x. PMID 10931172
- [Result] Merkus P, Guchelaar HJ, Bosch DA, Merkus FW. Direct access of drugs to the human brain after intranasal drug administration? Neurology. 2003 May 27;60(10):1669-71. doi: 10.1212/01.wnl.0000067993.60735.77. PMID 12771261
- [Result] Pearce RK, Owen A, Daniel S, Jenner P, Marsden CD. Alterations in the distribution of glutathione in the substantia nigra in Parkinson's disease. J Neural Transm (Vienna). 1997;104(6-7):661-77. doi: 10.1007/BF01291884. PMID 9444566
- [Result] Riederer P, Sofic E, Rausch WD, Schmidt B, Reynolds GP, Jellinger K, Youdim MB. Transition metals, ferritin, glutathione, and ascorbic acid in parkinsonian brains. J Neurochem. 1989 Feb;52(2):515-20. doi: 10.1111/j.1471-4159.1989.tb09150.x. PMID 2911028
- [Result] Sakhi AK, Russnes KM, Smeland S, Blomhoff R, Gundersen TE. Simultaneous quantification of reduced and oxidized glutathione in plasma using a two-dimensional chromatographic system with parallel porous graphitized carbon columns coupled with fluorescence and coulometric electrochemical detection. J Chromatogr A. 2006 Feb 3;1104(1-2):179-89. doi: 10.1016/j.chroma.2005.11.129. PMID 16376913
- [Result] Sechi G, Deledda MG, Bua G, Satta WM, Deiana GA, Pes GM, Rosati G. Reduced intravenous glutathione in the treatment of early Parkinson's disease. Prog Neuropsychopharmacol Biol Psychiatry. 1996 Oct;20(7):1159-70. doi: 10.1016/s0278-5846(96)00103-0. PMID 8938817
- [Result] Sian J, Dexter DT, Lees AJ, Daniel S, Agid Y, Javoy-Agid F, Jenner P, Marsden CD. Alterations in glutathione levels in Parkinson's disease and other neurodegenerative disorders affecting basal ganglia. Ann Neurol. 1994 Sep;36(3):348-55. doi: 10.1002/ana.410360305. PMID 8080242
- [Result] Sofic E, Lange KW, Jellinger K, Riederer P. Reduced and oxidized glutathione in the substantia nigra of patients with Parkinson's disease. Neurosci Lett. 1992 Aug 17;142(2):128-30. doi: 10.1016/0304-3940(92)90355-b. PMID 1454205
- [Result] Winter Y, Balzer-Geldsetzer M, Spottke A, Reese JP, Baum E, Klotsche J, Rieke J, Simonow A, Eggert K, Oertel WH, Dodel R. Longitudinal study of the socioeconomic burden of Parkinson's disease in Germany. Eur J Neurol. 2010 Sep;17(9):1156-1163. doi: 10.1111/j.1468-1331.2010.02984.x. Epub 2010 Mar 22. PMID 20345926
- [Result] Wolfe TR, Hillman TA, Bossart PJ. The comparative risks of bacterial contamination between a venturi atomizer and a positive displacement atomizer. Am J Rhinol. 2002 Jul-Aug;16(4):181-6; discussion 186. PMID 12222941